CLINICAL TRIAL: NCT02558569
Title: The Use of Fentanyl in General Anesthesia for Craniotomy With or Without 0.5% Levobupivacaine Scalp Block: A Randomized Controlled Trial
Brief Title: The Use of Fentanyl in General Anesthesia for Craniotomy With or Without 0.5% Levobupivacaine Scalp Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Manee Raksakietisak, Associate professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 359/2558(EC3
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Brain Tumor
Keywords: fentanyl, scalp block
MeSH Terms: conditions — Brain Neoplasms | interventions — Levobupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levobupivacaine (Experimental): Scalp nerve block with 0.5% Levobupivacaine adds up to intravenous fentanyl for intraoperative pain control during supratentorial craniotomy with brain tumor removal. The scalp block includes 4-6 nerves which give sensory supply to related location with the use of total 10-15 ml of 0.5% Levobupivacaine. Intravenous fentanyl is used for intraoperative analgesia in both groups with continuous infusion (1 mcg/kg/hr until opening of dura and then 0.5 mcg/kg/hr until finishing of dural closure) and increment doses (0.5 mcg/kg) also given. is used for intraoperative analgesia in both groups with continuous infusion (1 mcg/kg/hr until opening of dura and then 0.5 mcg/kg/hr until finishing of dural closure) and increment doses (0.5 mcg/kg) also given.
  Interventions: Drug: Levobupivacaine
- NSS (Sham Comparator): Scalp nerve block with 10-15 ml of 0.9% sodium chloride(NaCl), or normal saline (NSS) includes 4-6 nerves which give sensory supply to related location (sham block). Intravenous fentanyl is used for intraoperative analgesia in both groups with continuous infusion (1 mcg/kg/hr until opening of dura and then 0.5 mcg/kg/hr until finishing of dural closure) and increment doses (0.5 mcg/kg) also given.
  Interventions: Other: NSS

INTERVENTIONS:
Drug: Levobupivacaine — L form of bupivacaine with less cardiotoxicity.
  Other Names: Chirocaine
  Arms: Levobupivacaine
Other: NSS — Clear intravenous fluid looks alike local anesthetic.
  Other Names: 0.9% NaCl or Normal saline
  Arms: NSS

SUMMARY:
This study evaluates the use of fentanyl during craniotomy in two groups of brain tumor patients. The control group will receive standard general anesthesia with the use of fentanyl for intraoperative pain control and the study group will receive scalp nerve block with 0.5% levobupivacaine (local anesthetic) and also fentanyl for intraoperative pain control. The scalp nerve block might reduce the dose of fentanyl and promote faster emergence from general anesthesia.

DETAILED DESCRIPTION:
Fentanyl has widely been used for intraoperative analgesia for craniotomy. In craniotomy, the long and complex operation, the continuous infusion or repeated use of fentanyl can significantly delay emergence from general anesthesia. The scalp block with local anesthesia is widely used for awake craniotomy with great success but it is not routinely used in general craniotomy. In this study, the control group will receive standard general anesthesia with the use of fentanyl for intraoperative pain control and the study group will receive the addition of scalp nerve block with 0.5% levobupivacaine (local anesthetic). The scalp nerve block might reduce the total dose of fentanyl and promote faster emergence from general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* supratentorial brain tumor

Exclusion Criteria:

* tumor size>4 cm
* Glasgow Coma Score (GCS) <15
* already intubated
* uncontrolled hypertension
* can not communicate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The total dose of fentanyl being used during craniotomy | One day
  Total dose of fentanyl use during operative period

SECONDARY OUTCOMES:
Awakening time from general anesthesia | One day
  Time from the end of anesthetic to fully awake and extubation

CONTACTS AND LOCATIONS:
Overall Officials: Manee Raksakietisak, MD, Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Manee Raksakietisak, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok